CLINICAL TRIAL: NCT05158790
Title: Impact of Covid-19 on Training for Medical Residents Studying in ENT and Cervico-Facial Surgery Departments in France
Brief Title: Impact of Covid-19 on Training for ENT and Cervico-Facial Surgery Residents in France
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8476
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Cervico-Facial Surgery ENT Academic Medical and Surgical Training in France; Cervico-Facial Surgery ENT Medical Residency (Auvergne-Rhône-Alpes, Grand Est, Ile de France, Nouvelle Aquitaine and Provence-Alpes-Côte d'Azur Areas)
Keywords: Covid 19; Head and neck surgery; Residency; Medical training
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Administration of a questionnaire

SUMMARY:
The impact of the Covid-19 pandemic on medical education is real but little known.

ENT interns were directly affected by the management of Covid-19 patients (performing surgical tracheostomies), many conferences and trainings were cancelled, their usual hospital activity deeply reshuffled.

Although each student has a personal story of the impact of Covid-19 on their training, there is no doubt that the effects of Covid-19 are felt at scale. This study aims to investigate the effect of the pandemic on the medical and surgical training of ENT and Cervico-Facial Surgery interns in France from November 2019 to May 2021 (Auvergne-Rhône-Alpes, Grand Est, Ile de France, Nouvelle Aquitaine and Provence-Alpes-Côte d'Azur areas). A questionnaire will be sent by mail to ENT interns in France to assess the impact of Covid-19 on the training of ENT interns in France.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ENT residents in France (Auvergne-Rhône-Alpes, Grand Est, Ile de France, Nouvelle Aquitaine and Provence-Alpes-Côte d'Azur regions) during the period from November 2019 to May 2021.
* Informed of the objectives of the research and not objecting to the processing of their data

Exclusion Criteria:

- Subjects in research year, on availability, or in off-track training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ENT residents in France (Auvergne-Rhône-Alpes, Grand Est, Ile de France, Nouvelle Aquitaine and Provence-Alpes-Côte d'Azur regions) during the period from November 2019 to May 2021.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of Covid-19 on the training of ENT interns in France | before and during the acute phase of the pandemic from November 2019 to May 2021 (ordinal categorical primary endpoint)
  Evaluate the reduction in training time (practical and theoretical) as a proportion of usual training time between 2 periods: before and during the acute phase of the pandemic from November 2019 to May

SECONDARY OUTCOMES:
Assess interregional disparities in the impact of the Covid-19 crisis on ENT interns' training time. | before and during the acute phase of the pandemic, from November 2019 to May 2021
  Comparison of the reduction of time dedicated to training (practical and theoretical) between different regions of France. Percentage of time spent in the operating room, duty, on-call, DES course, IUD
  Comparison of the reduction of time dedicated to training (practical and theoretical) between different regions of France. Percentage of time spent in the operating room, duty, on-call, DES course, IUD.
Evaluate strategies implemented to compensate for block closure and theoretical course cancellations between waves | Before and during the acute phase of the pandemic, from November 2019 to May 2021
  Descriptive qualitative analysis of the strategies implemented.
Evaluate interregional disparities in training time for ENT interns outside the Covid-19 period. | Before and during the acute phase of the pandemic, from November 2019 to May 2021
  Comparison of the time dedicated to training (practical and theoretical) between different regions of France over a given period (pre-Covid19)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Service d'ORL et de Chirurgie Cervico-Faciale CHU Henri Mondor, APHP, Créteil
  - Service d'ORL et de Chirurgie Cervico-Faciale Hôpital Bicêtre, APHP, Le Kremlin-Bicêtre
  - Département d'ORL et de Chirurgie Cervico-Faciale Hôpital Gui de Chauliac, CHU de Montpellier, Montpellier
  - Service d'ORL et de Chirurgie Cervico-Faciale, Hôpital Lyon Sud, Pierre-Bénite
  - Service d'ORL et de Chirurgie Cervico-Faciale, CHU de Poitiers, Poitiers
  - Service d'ORL et de Chirurgie Cervico-Faciale Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No